CLINICAL TRIAL: NCT06656663
Title: INcreasing Adolescent Social and Community SupporT - Pilot
Acronym: INACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6735/017
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Loneliness
Keywords: Social Prescribing; Loneliness; School; Pupils; Link Worker

STUDY DESIGN:
Intervention Model Description: This study utilises a two-group (intervention vs. active control) parallel randomised design, with YP as the unit of randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Prescribing (Experimental): SP is a person-centred approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and Link Workers (LWs), based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have a good knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioural activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that best match their preferences.
  Interventions: Behavioral: Social Prescribing
- Signposting (Active Comparator): Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of school pastoral staff meeting with YP identified as lonely and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Interventions: Behavioral: Signposting

INTERVENTIONS:
Behavioral: Social Prescribing — SP is a person-centred approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and LW, based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have an excellent knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioural activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that best match their preferences.
  Arms: Social Prescribing
Behavioral: Signposting — Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of school pastoral staff meeting with YP identified as lonely and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Arms: Signposting

SUMMARY:
Background: Social prescribing is a mechanism of connecting patients with non-medical forms of support within the community and has been shown to improve loneliness. Yet uptake from young people has been lower than for adults. This is thought to be due to accessibility issues as young people are less likely to draw on primary care, where social prescribing in based, for wellbeing support. INACT will pilot a social prescribing pathway via schools to support young people who are lonely. It will test the feasibility and acceptability of delivering and evaluating it through a randomised controlled trial.

Methods: 78 pupils reporting loneliness will be recruited across 12 mainstream (6 primary and 6 secondary) schools in England and be randomly allocated to signposting or social prescribing. Pupils in the control group will receive signposting to sources of support from school staff. The co-produced social prescribing intervention includes up to 6 sessions with a Link Worker who will work with individuals to understand 'what matters to them' and connect them with local sources of support. Data will be collected at baseline, 3- and 6-months later. Acceptability and feasibility will be assessed via recruitment and retention, as well as via qualitative interviews. Interviews will also explore barriers, facilitators and mechanisms of change. Potential primary and secondary outcomes for a future trial will be completed to assess response and completeness, including measures of loneliness, mental health and wellbeing.

Discussion: INACT will provide preliminary evidence of the feasibility and acceptability of both the research design and social prescribing intervention. Results will inform a potential future randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people in a participating school and in Years 4, 5 or 7, 8
* Parental consent and young person assent is provided
* A score of 6 or above on the Good Childhood Index loneliness questions

Exclusion Criteria:

* Private schools
* Children and young people with severe learning disabilities

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | 3 Months
  Good Childhood Index is assessed using 3 questions on a 3-point Likert scale (scoring between 3-9). Higher scores indicate higher reported loneliness.
Intervention Feasibility (School Staff and Link Workers) | 6 months
  Feasibility of Intervention Measure (FIM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention feasibility
Intervention Acceptability (School Staff and Link Workers) | 6 months
  Acceptability of Intervention Measure (AIM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention acceptability
Intervention Appropriateness (School Staff and Link Workers) | 6 months
  Intervention Appropriateness Measure (IAM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention appropriateness

SECONDARY OUTCOMES:
Peer loneliness | 3 and 6 months
  LACA - Peer Subscale is assessed using 12 questions each on a four-point Likert scale (scoring between 12-48). Higher scores indicate higher peer loneliness
Wellbeing | 3 and 6 months
  Kidscreen-52 is assessed using 6 questions each on a five-point Likert scale (scoring between 6-30). Higher scores indicate greater well-being.
Mental health (emotional difficulties) | 3 and 6 months
  Me and My feelings is assessed using 10 questions on a 3-point Likert scale (scoring between 0-20). Higher scores indicate higher emotional difficulties
Service Use | 3 and 6 months
  Client Service Receipt of Inventory is assessed using 11 questions on a five-point Likert scale. Scoring can be looked at by individual items (i.e. score between 1-5) or by scoring all items (i.e. scores between 11-55). Higher scores indicate more contact with a service/services.
Stress | 3 and 6 months
  Perceived Stress Scale 4 is assessed using 4 questions on a five-point Likert scale (scoring between 0-16). Higher scores indicate higher levels of perceived stress
Loneliness | 6 Months
  Good Childhood Index is assessed using 3 questions on a three-point Likert scale (scoring between 3-9). Higher scores indicate higher reported loneliness.

OTHER OUTCOMES:
Family Support | Baseline only
  Moderator using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point likert scale (scoring between 4-20). Higher scores indicate higher family support.
School Support | Baseline only
  Moderator using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher school support.
Social support | 3 and 6 months
  Moderator using CYRM-R which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher social support
Local Environment | 3 and 6 months
  Moderator using questions from the HBSC 2022 assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate a more positive view of ones local environment
Activity Engagement | 3 and 6 months
  Moderator using questions from the BeeWell survey which is assessed using 11 questions each on a six-point Likert scale (scoring between 11-66). Higher scores indicate higher daily engagement with more activities. Each item can also be scored individually and indicates more frequent engagement with that activity.
Bullying | 3 and 6 months
  Moderator using kidscreen-52 (primary school pupils) which is assessed using 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher levels of bullying
Bullying | 3 and 6 months
  Moderator using the BeeWell survey (secondary school pupils) which is assessed using 3 questions each on a four-point Likert scale (scoring between 0-9). Higher scores indicate higher levels of bullying.
Social structure and quality | 3 and 6 months
  Moderator using questions adapted from PISA 2022 and MCS4 which is assessed using five questions. One of which requires an open-ended numerical value and four questions which are rated on a five-point Likert scale (scoring between 0-16). Higher scores indicate a greater social structure and friendship quality.
Problem Solving | 3 and 6 months
  Mechanism using the Student Resilience Survey which is assessed using 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher problem solving with others
Flow | 3 and 6 months
  Mechanism using the General Flow Proneness Scale (secondary school pupils only) which is assessed using 13 questions each on a five-point Likert scale (scoring between 13-65). Higher scores indicate higher flow experience
Therapeutic Alliance | 3 and 6 months
  Mechanism using the Session Feedback Questionnaire which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher therapeutic alliance. This is for individuals in the social prescribing intervention only

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Some IPD data will be shared but we specific data is being currently discussed with the funder. We will update this record when we know more.

REFERENCES:
- [Derived] Hayes D, Burton A, Bu F, Humphrey N, Qualter P, Han E, Sticpewich L, Wright J, Bone JK, Maguire S, Gonzalez Umpierrez LC, Stapley E, Tibber MS, Fancourt D. INcreasing Adolescent social and Community supporT (INACT): Pilot study protocol. PLoS One. 2025 Mar 26;20(3):e0317823. doi: 10.1371/journal.pone.0317823. eCollection 2025. PMID 40138284
- See also: Study webpage overview — https://sbbresearch.org/projects/inact-increasing-adolescent-social-and-community-support/